CLINICAL TRIAL: NCT00193466
Title: Phase II Trial of Rituximab/Fludarabine Followed by CAMPATH-1H in the First-Line Treatment of Patients With Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL)
Brief Title: Rituximab and Fludarabine Followed by CAMPATH-1H in Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Bayer (Industry)
Responsible Party: John D. Hainsworth, M.D., Sarah Cannon Research Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LYM 21; CAM-217
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2010-12-30 (Estimated); Status verified 2010-12

CONDITIONS: Non-Hodgkins Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab; fludarabine

INTERVENTIONS:
Drug: Rituximab
Drug: Fludarabine
Drug: CAMPTH-1H

SUMMARY:
In this multicenter trial, we will investigate the use of fludarabine plus rituximab, followed by Campath-1H, in previously untreated patients with CLL/SLL. Patients who are elderly, or who are considered unlikely to tolerate this combination therapy well, will receive single agent rituximab followed by Campath-1H.

DETAILED DESCRIPTION:
Upon determination of eligibility, all patients will receive:

Fludarabine + Rituximab + CAMPATH-1H

Patients who are judged by the investigator not to be candidates for fludarabine due to advanced age, marginal performance status or coexistent medical conditions will receive rituximab alone followed by CAMPATH-1H.

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Histologically proven B-cell CLL/SLL
* Positive staining for CD20 antigen
* No systemic chemotherapy.
* Measurable or evaluable disease
* Able to perform activities of daily living with minimal assistance
* Age > 18 years
* Life expectancy > 12 weeks
* Adequate liver and kidney function
* Must be accessible for treatment and follow-up
* Must give written informed consent prior to entering this study.

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Female pregnant or lactating
* Unstabilized active infection on the basis of neutropenia
* History of previous severe opportunistic infections
* Serious underlying medical conditions
* Central nervous system involvement
* History of other neoplasms, either active or treated within five years

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2002-01; Primary Completion 2007-01 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Complete response rate

SECONDARY OUTCOMES:
Molecular complete response rate
Progression free survival
Overall toxicity

CONTACTS AND LOCATIONS:
Overall Officials: John D. Hainsworth, MD, Principal Investigator — SCRI Development Innovations, LLC

REFERENCES:
- [Result] Hainsworth JD, Vazquez ER, Spigel DR, Raefsky E, Bearden JD, Saez RA, Greco FA. Combination therapy with fludarabine and rituximab followed by alemtuzumab in the first-line treatment of patients with chronic lymphocytic leukemia or small lymphocytic lymphoma: a phase 2 trial of the Minnie Pearl Cancer Research Network. Cancer. 2008 Mar 15;112(6):1288-95. doi: 10.1002/cncr.23271. PMID 18189296